CLINICAL TRIAL: NCT02512250
Title: Swiss Hemophilia Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Swiss Hemophilia Network (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-0667
Record Dates: First submitted 2015-07-26; First posted 2015-07-30 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Hemophilia and Other Severe Bleeding Disorders
MeSH Terms: conditions — Hemophilia A | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Registry

SUMMARY:
The Swiss Hemophilia Registry will collect data on the prophylactic and therapeutic use of factor concentrates in patients with hemophilia and other severe bleeding disorders in Switzerland.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of hemophilia or other severe bleeding disorders. Signed inform consent

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hemophilia and other severe bleeding disorders
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2015-05; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of incidence of disease and inhibitor development | 1 year
  Demographics, Comorbidties, factor consumption for prophylaxis, bleeding and surgery, inhibito develeopment

CONTACTS AND LOCATIONS:
Locations (19):
- Switzerland (19):
  - Kantonsspital Aarau Zentrum für Onkologie/Hämatologie und Transfusionsmedizin, Aarau
  - Kinderklinik, Aarau
  - Universitätsspital Basel Diagnostische Hämatologie, Basel
  - Universitätskinderspital beider Basel (UKBB) Abteilung Onkologie/Hämatologie, Basel
  - Ospedale San Giovanni, Bellinzona
  - Servizio di Ematologia Ospedale Regionale di Bellinzona e Valli, Bellinzona
  - Inselspital, Universitätsspital Bern Poliklinik für Hämatologie, Bern
  - Kantonspital Graubünden, Chur
  - Unité d'Hémostase HUG, Geneva
  - Unité d'Oncologie-Hématologie pédiatrique, Hôpital des Enfants HUG, Geneva
  - Centre Hospitalier Universitaire Vaudois Service d'Hématologie, Lausanne
  - Policlinique d'onco-hématologie péd., CHUV, Lausanne
  - Kantonsspital Luzern Abteilung Hämatologie, Lucerne
  - Kinderspital Luzern, Lucerne
  - Ostschweizer Kinderspital St. Gallen, Sankt Gallen
  - Kantonspital St. Gallen, Sankt Gallen
  - Kinder und Erwachsenenzentrum Sion Service Régional Valaisan de Transfusion Sanguine CRS, Sion
  - University Children's Hospital, Zurich
  - University Hospital Zürich, Zurich